CLINICAL TRIAL: NCT01083732
Title: Single Dose Open-label PK/PD, Safety and Tolerability Study of Dabigatran Etexilate Mesilate Given at the End of Standard Anticoagulant Therapy in Successive Groups of Children Aged 2 Years to Less Than 12 Years Followed by 1 Year to Less Than 2 Years
Brief Title: Safety and Tolerability of Dabigatran Etexilate Solution in Children 1 to < 12 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1160.89; 2009-013618-29 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

ARMS (1):
- dabigatran etexilate (Experimental): treatment with dabigatran oral solution as a single dose
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — Experimental dose chosen based on age and weight

SUMMARY:
To investigate the safety and tolerability of dabigatran etexilate solution in children and to obtain preliminary pharmacokinetic/pharmacodynamic data

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

1. males or females 1 to less than 12 years of age
2. objective diagnosis of primary VTE
3. completion of planned treatment course with LMWH or OAC for primary VTE
4. written informed consent by parent (legal guardian) and patient assent (if applicable)

Exclusion criteria:

1. weight less than 9 kg
2. conditions associated with increased risk of bleeding
3. patients who have any condition that would not allow safe participation in study Note: Further exclusion criteria apply

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2010-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Boehringer Ingelheim Investigational Site, Ottawa, Ontario, Canada
- Boehringer Ingelheim Investigational Site, Roma, Italy
- Boehringer Ingelheim Investigational Site, Vilnius, Lithuania
- Boehringer Ingelheim Investigational Site, Kazan', Russia
- Boehringer Ingelheim Investigational Site, Zurich, Switzerland
- Thailand (2):
  - Boehringer Ingelheim Investigational Site, Bangkok
  - Boehringer Ingelheim Investigational Site, Khon Kaen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients were enrolled, 18 patients were entered and treated, 2 patients were screening failures.
Pre-assignment Details: Open-label, multicentre, non-randomised, uncontrolled, single arm study.
Groups:
- Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years):: The patients aged 1 to <2 years were orally administered a single dose of dabigatran etexilate (Dabigatran etexilate oral liquid formulation (6.25 mg/mL) after reconstitution from dabigatran etexilate granules (167.5 mg) and solvent for oral liquid formulation)
- Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years): The patients aged 2 to <12 years were orally administered a single dose of dabigatran etexilate (Dabigatran etexilate oral liquid formulation (6.25 mg/mL) after reconstitution from dabigatran etexilate granules (167.5 mg) and solvent for oral liquid formulation)
- Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years): The patients aged 2 to <12 years were orally administered a multiple dose (3 days, twice daily) of dabigatran etexilate (Dabigatran etexilate oral liquid formulation (6.25 mg/mL) after reconstitution from dabigatran etexilate granules (167.5 mg) and solvent for oral liquid formulation)
Period: Overall Study
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years): | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Started | 6 | 9 | 3
Completed | 6 | 9 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all subjects who were dispensed study medication and were documented to have taken at least 1 dose of trial medication.
Groups:
- Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years): The patients aged 1 to <2 years were orally administered a single dose of dabigatran etexilate (Dabigatran etexilate oral liquid formulation (6.25 mg/mL) after reconstitution from dabigatran etexilate granules (167.5 mg) and solvent for oral liquid formulation)
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years) | Total
Number analyzed (Participants) | 6 | 9 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.0 (0.0) | 5.2 (2.6) | 8.3 (2.5) | 4.3 (3.3)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 4 | 6 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Total Dabigatran (SUM BIBR 953 ZW)
Description: Plasma concentration of total dabigatran (SUM BIBR 953 ZW)
Time Frame: At 1 hour (h), 2 h, 4 h, 6 h, and 10 h after single administration of dabigatran etexilate and at 2 h, 50 h, and 72 h after multiple dose administration of dabigatran etexilate
Population: Pharmacokinetic set (PKS): This patient set included all treated patients who provided at least one pharmacokinetic/ pharmacodynamic (PK/PD) observation and had no important protocol violations (PVs) with respect to the statistical analysis of PK or PD endpoints.
  PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9 | 3
ng/mL
  1h (N= 4, 9, NA) | 79.4 (45.6) | 90.6 (48.8) | NA (NA) — Time-point is not applicable for multiple dose group
  2h (N=6, 9, 2) | 129.0 (9.84) | 114.0 (37.9) | 26.0 (62.6)
  4h (N=6, 9, NA) | 91.0 (23.0) | 87.7 (31.6) | NA (NA) — Time-point is not applicable for multiple dose group
  6h (N=6, 9, NA) | 62.9 (32.6) | 56.2 (34.2) | NA (NA) — Time-point is not applicable for multiple dose group
  10h (N=6, 9, NA) | 34.8 (41.4) | 28.2 (37.0) | NA (NA) — Time-point is not applicable for multiple dose group
  50h (N=NA, NA, 2) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Time-point is not applicable for single dose group | 46.0 (64.7)
  72h (N=NA, NA, 3) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Time-point is not applicable for single dose group | 11.9 (47.8)

2. Primary Outcome: Plasma Concentration of Free Dabigatran (BIBR 953 ZW).
Description: Plasma concentration of free dabigatran (BIBR 953 ZW)
Time Frame: as for outcome 1
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9 | 3
ng/mL
  1h (N= 4, 9, NA) | 68.5 (43.8) | 80.0 (43.9) | NA (NA) — Time-point is not applicable for multiple dose group
  2h (N=6, 9, 2) | 101.0 (12.8) | 98.5 (35.3) | 23.4 (72.2)
  4h (N=6, 9, NA) | 75.3 (30.2) | 74.5 (31.7) | NA (NA) — Time-point is not applicable for multiple dose group
  6h (N=6, 9, NA) | 51.6 (40.0) | 48.4 (37.9) | NA (NA) — Time-point is not applicable for multiple dose group
  10h (N=6, 9, NA) | 28.1 (49.8) | 23.7 (40.3) | NA (NA) — Time-point is not applicable for multiple dose group
  50h (N=NA, NA, 2) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Time-point is not applicable for single dose group | 37.3 (60.7)
  72h (N=NA, NA, 3) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Time-point is not applicable for single dose group | 8.43 (44.0)

3. Primary Outcome: Plasma Concentration of Unchanged Dabigatran Etexilate (BIBR 1048 BS)
Description: Plasma concentration of unchanged dabigatran etexilate (BIBR 1048 BS).
  Some values are "NA" because Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the Geometric Mean (gMean) and Geometric Coefficient of Variation (gCV) is not calculated according to internal rules.
Time Frame: as for outcome 1
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Dabigatran Etexilate (Single Dose, Age Group 1 to <12 Years): The patients aged 1 to <12 years were orally administered a single dose of dabigatran etexilate (Dabigatran etexilate oral liquid formulation (6.25 mg/mL) after reconstitution from dabigatran etexilate granules (167.5 mg) and solvent for oral liquid formulation)
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 15 | 3
ng/mL
  1h (N= 13, NA) | 3.82 (107) | NA (NA) — Time-point is not applicable for multiple dose group
  2h (N=5, 2) | 3.23 (74.4) | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules
  4h (N=15, NA) | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules | NA (NA) — Time-point is not applicable for multiple dose group
  6h (N=1, NA) | 1.05 (NA) — All patients except one patient had values below the limit of quantification. | NA (NA) — Time-point is not applicable for multiple dose group
  10h (N=15, NA) | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules | NA (NA) — Time-point is not applicable for multiple dose group
  50h (N=NA, 2) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules
  72h (N=NA, 3) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules

4. Primary Outcome: Plasma Concentration of Metabolite BIBR 951 BS
Description: Plasma concentration of metabolite BIBR 951 BS
Time Frame: as for outcome 1
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 15 | 3
ng/mL
  1h (N=13, NA) | 4.88 (82.2) | NA (NA) — Time-point is not applicable for multiple dose group
  2h (N=15, 2) | 3.55 (83.0) | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules
  4h (N=4, NA) | 1.71 (52.8) | NA (NA) — Time-point is not applicable for multiple dose group
  6h (N=15, NA) | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules | NA (NA) — Time-point is not applicable for multiple dose group
  10h (N=15, NA) | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules | NA (NA) — Time-point is not applicable for multiple dose group
  50h (N=NA, 2) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules
  72h (N=NA, 3) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Values were below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules

5. Primary Outcome: Plasma Concentration of Metabolite BIBR 1087 SE
Description: Plasma concentration of metabolite BIBR 1087 SE
Time Frame: as for outcome 1
Population: Pharmacokinetic set (PKS): This patient set included all treated patients who provided at least one pharmacokinetic/ pharmacodynamic (PK/PD) observation and had no important protocol violations (PVs) with respect to the statistical analysis of PK or PD endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 15 | 3
ng/mL
  1h (N=12, NA) | 2.31 (54.0) | NA (NA) — Time-point is not applicable for multiple dose group
  2h (N=8, 2) | 1.51 (38.5) | NA (NA) — Values below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.
  4h (N=1, NA) | 1.18 (NA) — All patients except one patient had values below the limit of quantification. | NA (NA) — Time-point is not applicable for multiple dose group
  6h (N=15, NA) | NA (NA) — Values below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | NA (NA) — Time-point is not applicable for multiple dose group
  10h (N=15, NA) | NA (NA) — Values below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | NA (NA) — Time-point is not applicable for multiple dose group
  50h (N=NA, 2) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Values below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.
  72h (N=NA, 3) | NA (NA) — Time-point is not applicable for single dose group | NA (NA) — Values below the limit of quantification. Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

6. Primary Outcome: Central Measurement of Activated Partial Thromboplastin Time (aPTT) at Predose and 2 and 10 h After Intake of Study Medication.
Description: Central measurement of aPTT (activated partial thromboplastin time) at predose and 2 and 10 h after intake of study medication. For multiple dose patients only local measurements were planned. The Standard Deviation presented below is actually the % coefficient of variation.
Time Frame: at predose and 2 and 10 h after intake of study medication.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9
seconds
  Ebase (N=6, 7) | 32.3 (24.6) | 34.9 (24.5)
  E2 (N=6, 9) | 47.5 (24.7) | 77.0 (54.6)
  E10 (N=5, 8) | 40.3 (19.6) | 58.4 (40.6)

7. Primary Outcome: Central Measurement of Ecarin Clotting Time (ECT) at Predose and 2 and 10 h After Intake of Study Medication.
Description: Central measurement of ECT (ecarin clotting time) at predose and 2 and 10 h after intake of study medication. ECT was not planned to be measured in the multiple dose group. The Standard Deviation presented below are actually the % coefficient of variation
Time Frame: at predose and 2 and 10 h after intake of study medication.
Population: PKS (evaluable cases)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9
seconds
  Ebase (N=6, 6) | 36.9 (7.49) | 36.8 (10.5)
  E2 (N=6, 7) | 79.8 (5.15) | 73.6 (22.1)
  E10 (N=5, 7) | 49.7 (5.36) | 52.2 (10.3)

8. Primary Outcome: Central Measurement of Diluted Thrombin Time (dTT) at Predose and 2 and 10 h After Intake of Study Medication.
Description: Central measurement of dTT (diluted thrombin time) at predose and 2 and 10 h after intake of study medication. The Standard Deviation presented below are actually the % coefficient of variation
Time Frame: at predose and 2 and 10 h after intake of study medication.
Population: PKS (evaluable cases)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9 | 3
seconds
  Ebase (N=6, 9, 2) | 31.9 (4.67) | 35.6 (10.1) | 32.9 (4.73)
  E2 (N=6, 9, 2) | 46.6 (6.02) | 53.6 (18.4) | 34.3 (1.24)
  E10 (N=6, 9, NA) | 35.5 (6.02) | 39.7 (9.76) | NA (NA) — Time-point is not applicable for multiple dose group

9. Primary Outcome: Cmax (Maximum Measured Concentration of Total Dabigatran in Plasma)
Description: Cmax (maximum measured concentration of total dabigatran in plasma). Endpoint can only be calculated for single dose patients. For multiple dose patients the time points do not allow calculation of Cmax (no profile, only one measurement after selected doses, refer to primary outcome no. 1 and 2).
Time Frame: At 1 hour (h), 2 h, 4 h, 6 h, and 10 h after single administration of dabigatran etexilate
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9
ng/mL | 129 (9.84) | 116 (38.6)

10. Primary Outcome: Tmax (Time From Dosing to Maximum Measured Concentration of Total Dabigatran in Plasma)
Description: tmax (time from dosing to maximum measured concentration of total dabigatran in plasma).
  Endpoint can only be calculated for single dose patients. For multiple dose patients the time points do not allow calculation of tmax (no profile, only one measurement after selected doses, refer to primary outcome no. 1 and 2).
Time Frame: At 1 hour (h), 2 h, 4 h, 6 h, and 10 h after single administration of dabigatran etexilate
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9
hours | 1.99 (9.84) [1.92 to 2.20] | 2.00 (38.6) [1.03 to 4.02]

11. Primary Outcome: AUC0-tz (Area Under the Concentration Time Curve of the Total Dabigatran in Plasma Over the Time Interval 0 up to the Last Quantifiable Data Point)
Description: AUC0-tz (area under the concentration time curve of the total dabigatran in plasma over the time interval 0 up to the last quantifiable data point).
  Endpoint can only be calculated for single dose patients. For multiple dose patients the time points do not allow calculation of AUC0-tz (no profile, only one measurement after selected doses, refer to primary outcome no. 1 and 2).
Time Frame: At 1 hour (h), 2 h, 4 h, 6 h, and 10 h after single administration of dabigatran etexilate
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9
ng*h/mL | 715 (22.5) | 658 (32.5)

12. Primary Outcome: Cmax (Maximum Measured Concentration of Free Dabigatran in Plasma)
Description: Cmax (maximum measured concentration of free dabigatran in plasma). Endpoint can only be calculated for single dose patients. For multiple dose patients the time points do not allow calculation of Cmax (no profile, only one measurement after selected doses, refer to primary outcome no. 1 and 2).
Time Frame: At 1 hour (h), 2 h, 4 h, 6 h, and 10 h after single administration of dabigatran etexilate
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9
ng/mL | 101 (12.8) | 102 (36.9)

13. Primary Outcome: Tmax (Time From Dosing to Maximum Measured Concentration of Free Dabigatran in Plasma)
Description: tmax (time from dosing to maximum measured concentration of free dabigatran in plasma).
  Endpoint can only be calculated for single dose patients. For multiple dose patients the time points do not allow calculation of tmax (no profile, only one measurement after selected doses, refer to primary outcome no. 1 and 2).
Time Frame: At 1 hour (h), 2 h, 4 h, 6 h, and 10 h after single administration of dabigatran etexilate
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9
hours | 1.99 (9.84) [1.92 to 2.20] | 2.00 (38.6) [1.08 to 2.08]

14. Primary Outcome: AUC0-tz (Area Under the Concentration Time Curve of the Free Dabigatran in Plasma Over the Time Interval 0 up to the Last Quantifiable Data Point)
Description: AUC0-tz (area under the concentration time curve of the free dabigatran in plasma over the time interval 0 up to the last quantifiable data point).
  Endpoint can only be calculated for single dose patients. For multiple dose patients the time points do not allow calculation of AUC0-tz (no profile, only one measurement after selected doses, refer to primary outcome no. 1 and 2).
Time Frame: At 1 hour (h), 2 h, 4 h, 6 h, and 10 h after single administration of dabigatran etexilate
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9
ng*h/mL | 581 (27.7) | 566 (32.2)

15. Primary Outcome: Percentage of Patients With Incidence of Any Bleeding Events (Major, Clinically Relevant Non-major (CRNM) and Minor) During the Treatment Period.
Description: Major: Fatal bleeding, Clinically overt bleeding associated with decrease in haemoglobin of at least 2 g/dL in 24-h-period,bleeding that was retroperitoneal,pulmonary,intracranial,or otherwise involved the central nervous system,bleeding that required surgical intervention in an operating suite. CRNM: Overt bleeding for which a blood product was administered & which was not directly attributable to the patient's underlying medical condition,bleeding that required medical or surgical intervention to restore haemostasis,other than in an operating suite. Minor: Any overt or macroscopic evidence of bleeding that did not fulfil the criteria for either major bleeding or CRNM bleeding. For multiple dosing,all events with an onset date after the date of first dose until the end of trial treatment including 3 days after the last treatment and for single dosing,all events with an onset during the 48-h-period after study medication intake were assigned to the on-treatment period.
Time Frame: Up to 6 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9 | 3
Percentage of participants | 0.0 (22.5) | 0.0 (32.5) | 0.0

16. Secondary Outcome: Percentage of Patients With Any Adverse Events During the Treatment Period
Description: Percentage of patients with any adverse events during the treatment period. For patients with multiple dosing, all AEs with an onset date after the date of first dose until the end of trial treatment including 3 days after the last treatment were assigned to the on-treatment period. For patients with single dosing, all AEs with an onset during the 48-h-period after study medication intake were assigned to the on-treatment period.
Time Frame: Up to 6 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9 | 3
Percentage of participants | 0.0 (22.5) | 0.0 (32.5) | 33.3

17. Secondary Outcome: Global Assessment of Tolerability of Study Medication- Taste Assessment
Description: The investigator was to provide a global clinical assessment of tolerability including patient taste assessment.This assessment was based on 6-point scale (Very good, good, satisfactory, bad, very bad, missing). The taste assessment was only provided when the patient was old enough to evaluate the taste.
Time Frame: Day 1 (immediately after dosing)
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9 | 3
Percentage of participants
  Very Good | 0 (22.5) | 0 (32.5) | 0
  Good | 0 | 0 | 0
  Satisfactory | 0 | 44.44 | 33.33
  Bad | 0 | 0 | 66.67
  Very Bad | 0 | 33.33 | 0
  Missing | 100.00 | 22.22 | 0

18. Secondary Outcome: Percentage of Patients With Changes in Laboratory and Clinical Parameters Such as Liver Enzymes and Physical Examination
Description: Percentage of patients with changes in laboratory and clinical parameters such as liver enzymes and physical examination.
  Clinically Relevant Abnormalities for Laboratory Parameters were reported.
Time Frame: During the treatment period, Up to 6 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9 | 3
Percentage of participants | 0.0 (22.5) | 0.0 (32.5) | 0.0

19. Secondary Outcome: Global Assessment of Tolerability of Study Medication
Description: The investigator was to provide a global clinical assessment of tolerability of study medication by the patient.This assessment was based on 5-point scale (good, satisfactory, not satisfactory, bad, not assessable).
Time Frame: Day 1 (immediately after dosing)
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Number analyzed (Participants) | 6 | 9 | 3
Percentage of participants
  Good | 33.33 (22.5) | 11.11 (32.5) | 100.00
  Satisfactory | 16.67 | 22.22 | 0
  Not satisfactory | 33.33 | 44.44 | 0
  Bad | 0 | 22.22 | 0
  Not assessable | 16.67 | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) during the treatment period, up to 6 days.
Description: For patients with multiple dosing, all AEs with an onset date after the date of first dose until the end of trial treatment including 3 days after the last treatment and for patients with single dosing, all AEs with an onset during the 48-h-period after study medication intake were assigned to the on-treatment period.
Arm/Group | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (Single Dose, Age Group 1 to <2 Years) (N=6) | Dabigatran Etexilate (Single Dose, Age Group 2 to <12 Years) (N=9) | Dabigatran Etexilate (Multiple Dose, Age Group 2 to <12 Years) (N=3)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights